CLINICAL TRIAL: NCT03222050
Title: Effectiveness of Distraction Techniques on Pain Intensity During Immunization Among Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Preeti dabas, Student, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 777
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- electronic toy group (Experimental): Distraction technique was given by electronic toy during immunization and started 30 seconds before immunization and it lasted until 15 seconds
  Interventions: Other: Distraction technique
- key toy group (Experimental): Distraction technique was given by key toy during immunization and started 30 seconds before immunization and it lasted until 15 seconds
  Interventions: Other: Distraction technique
- Simple toy group (Experimental): Distraction technique was given by simple toy during immunization and started 30 seconds before immunization and it lasted until 15 seconds
  Interventions: Other: Distraction technique
- control group (No Intervention): Routine care was given during immunization and no intervention was given

INTERVENTIONS:
Other: Distraction technique
  Arms: Simple toy group; electronic toy group; key toy group

SUMMARY:
A study to assess and compare the effectiveness of Distraction techniques on Pain intensity during Immunization among Infants in selected hospital of Ambala, Haryana.

DETAILED DESCRIPTION:
Immunization is an important part of public health intervention and cost effective strategy to control the infectious diseases especially in children and it is one of the most common painful procedure in infants. Pain during immunization leads to distressing experience for the infant, parents and health care worker. Distraction is non pharmacological method which is used for diverting attention from noxious stimulus by passively redirecting the attention or by actively performed by the subject in the performance of diversion technique. Aim and objectives:The aim of present study was to compare the effectiveness of distraction techniques on pain intensity during immunization among infants. The objectives of the study were to assess and compare the mean pain scores among infants receiving immunization in electronic toy group, key toy group, simple toy group and control group and to find out the association of pain scores among infants receiving immunization with their selected variables. Material and methods: A true experimental multiple intervention post test control design was used. There were 100 infants selected using simple random sampling technique and were randomly allocated in various groups such as electronic toy group, key toy group, simple toy group and control group using lottery method. During immunization, distraction techniques were shown to experimental groups and routine care was given to control group. Research tool was submitted to 7 experts from various specialists for validity. Reliability was calculated by Kappa method and it was 0.83 of FLACC pain scale to assess pain intensity during immunization among infants. Data collection was done in January 2017. The obtained data was analyzed and interpreted in terms of objectives and research hypotheses. Analysis was done by using descriptive and inferential statistics.

ELIGIBILITY:
Inclusion Criteria:

* • Infants who were-visiting immunization clinics of Civil Hospital for immunization.

having 10 and 14 weeks of age. receiving pentavalent vaccine. Parents and caregivers who were willing to give consent

Exclusion Criteria:

The study excluded infants who: had undergone any painful procedure 2 hour prior to immunization, were visually or hearing disabled.

had history of seizures, use of topical anesthetics at immunization site, use of sedatives, analgesics or opioids in the preceding 24 hours.

Ages: 10 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Flacc pain score | 5 minute
  Flacc pain score
  Level of pain:
  0 - No distress/Pain 1-3 - Mild distress/Pain 4-7 - Moderate distress/Pain 8-10 - Severe distress/Pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Hockenberry Marilyn. Wong's Essentials of Pediatric Nursing. 7th Edition. New Delhi. Elsevier Publication (P) Ltd. 2007; 235-238.
- [Background] 2. Wong DL, Hocken MJ. Nursing care of infants and children and adolescents. Agency for Healthcare Policy and Research Publication. 1992.
- [Result] 9. Sharma Rimple, Kaur Charanjit. A Randomized control trial to assess the effect of distraction technique on pain during immunization among infants. International journal of current research. June 2014:6:7119-7123.